CLINICAL TRIAL: NCT00693966
Title: A Phase II Double-Blind, Randomized, Dose-Comparison Study to Evaluate the Safety and Immunogenicity of MEDI-517, a Virus-Like Particle Vaccine Against Human Papillomavirus Types 16 and 18, in Healthy Adult Female Volunteers
Brief Title: Dose-Comparison Study to Evaluate the Safety and Immunogenicity of MEDI-517 (GSK 580299) in Healthy Adult Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 580299/005
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Papillomavirus
Keywords: HPV, Vaccine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Formulation 1 of the vaccine (MEDI-517 HPV-16/18 VLP AS04 vaccine)
  Interventions: Biological: MEDI-517 HPV-16/18 VLP AS04 vaccine (Formulation 1)
- Group B (Experimental): Formulation 2 of the vaccine
  Interventions: Biological: MEDI-517 HPV-16/18 VLP AS04 vaccine (Formulation 2)
- Group C (Experimental): Formulation 3 of the vaccine
  Interventions: Biological: MEDI-517 HPV-16/18 VLP AS04 vaccine (Formulation 3)
- Group D (Experimental): Formulation 4 of the vaccine [with Al(OH)3]
  Interventions: Biological: MEDI-517 HPV-16/18 VLP with Al(OH)3 (Formulation 4)

INTERVENTIONS:
Biological: MEDI-517 HPV-16/18 VLP AS04 vaccine (Formulation 1) — IM injection
  Arms: Group A
Biological: MEDI-517 HPV-16/18 VLP AS04 vaccine (Formulation 2) — IM injection
  Arms: Group B
Biological: MEDI-517 HPV-16/18 VLP AS04 vaccine (Formulation 3) — IM injection
  Arms: Group C
Biological: MEDI-517 HPV-16/18 VLP with Al(OH)3 (Formulation 4) — IM injection
  Other Names: MEDI-517 HPV-16/18 VLP AS04 vaccine (Formulation 2); MEDI-517 HPV-16/18 VLP AS04 vaccine (Formulation 3); MEDI-517 HPV-16/18 VLP AS04 vaccine (Formulation 1)
  Arms: Group D

SUMMARY:
The purpose of this Phase II study is to provide data regarding the safety and immunogenicity for a range of dose levels of MEDI-517 in women who are HPV-16/18 seronegative and negative for high-risk HPV DNA. The study is designed to evaluate safety and immunogenicity data for MEDI-517 when formulated with either AS04 or aluminum hydroxide. Extended follow-up will provide long-term immune response data.

This study was originally performed by MedImmune. However, GSK is now responsible for the clinical development of the HPV vaccine.

DETAILED DESCRIPTION:
This is a Phase II double-blind, randomized, dose-comparison, multicenter study in the United States of three different dose levels of MEDI-517 (HPV-16/18 VLP AS04 vaccine) and one dose of MEDI-517 formulated with aluminum hydroxide, with doses administered at 0, 30 and 180 days. Healthy female volunteers 18 through 30 years of age will be entered into 4 treatment arms. The objectives of study are to evaluate reactogenicity, safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 through 30 years of age (must not have reached the 31st birthday)
* Unless previously surgically sterilized, agrees to use an effective method of birth control beginning 30 days before the first study injection and continuing through 60 days after the final study injection
* Healthy by medical history and physical examination
* Seronegative for HPV-16 and HPV-18 antibody by ELISA within 21 days of study entry
* Cervical specimen negative for high-risk HPV DNA using the Digene Hybrid Capture® II HPV test (high-risk types Probe B) within 21 days of study entry
* Normal Pap smear, using the Cytyc ThinPrep® Pap Test, within 21 days of study entry
* No evidence of anogenital HPV lesions or no physical findings suggestive of other gynecologic pathogens on pelvic examination within 21 days of study entry
* Agrees to no other experimental therapy or vaccines until 30 days after the last study injection
* Written informed consent obtained from the volunteer

Exclusion Criteria:

* Acute illness or fever (oral temperature ≥ 99.5°F [37.5°C]) at start of the study
* History or clinical manifestations of significant medical or psychiatric disorder
* Pregnant or lactating
* Use of immunosuppressive medication within the previous 90 days or history of immunodeficiency
* History of cancer
* History of alcohol or drug abuse within the past 2 years
* Abnormal laboratory values in the screening panel which in the opinion of the principal investigator are judged to be clinically significant
* Receipt of immunoglobulin or blood products within 90 days prior to study entry
* History of abnormal Pap smear (other than a single prior report of ASCUS or indeterminate Pap smear with a subsequent normal report)
* Positive tests for hepatitis C antibody, hepatitis B surface antigen, or HIV-1 antibody
* Any prior receipt of any vaccine (experimental or otherwise) for treatment or prophylaxis of genital warts or other papillomavirus related condition. Any treatment of genital warts or other papillomavirus related condition within 6 months of randomization (local therapy for common skin and/or plantar warts is allowed)
* Previous administration of any components of the investigational vaccine
* Receipt of any experimental vaccine within 90 days prior to entry into this study
* Receipt of any experimental drug therapy within 30 days or five half-lives of the experimental drug (if the half-life is known), whichever is longer

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 1999-10; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Solicited adverse event rates (including injection site and systemic reactions) | For 7 days after each injection
Unsolicited adverse event rates | For 30 days after each injection
Serious adverse event rates | From first injection through 30 days after last injection
Laboratory assessments (Biochemistry and Hematology parameters) | Study Days 0, 30 and 210
Vital signs (temperature, blood pressure, pulse rate, respiratory rate) | At the time of injection and 30 minutes after the injection
Serum ELISA titers against HPV-16 and HPV-18 | 30 days after the third injection

SECONDARY OUTCOMES:
Serum ELISA titers against HPV-16 and HPV-18 | Study Days 0, 7, 30, 60, 180, 210, and 360, and at 24, 36, and 48 months
Neutralization titers against HPV-16 and HPV-18 | Study Days 0, 60, 210 and 360
Cell-mediated immunity by IL-5, IFN-γ and lymphoproliferative assays | Study Days 0, 60, 210, and 360
HPV-16 and HPV-18 ELISA and inhibitory ELISA | Study Days 0, 60, 210, and 360, and at 18, 24, 36, and 48 months
Cervical and vaginal ELISA titers against HPV-16 and HPV-18 | At Study Days 210 and 360

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Descamps D, Hardt K, Spiessens B, Izurieta P, Verstraeten T, Breuer T, Dubin G. Safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine for cervical cancer prevention: a pooled analysis of 11 clinical trials. Hum Vaccin. 2009 May;5(5):332-40. doi: 10.4161/hv.5.5.7211. Epub 2009 May 20. PMID 19221517
- [Background] Giannini SL, Hanon E, Moris P, Van Mechelen M, Morel S, Dessy F, Fourneau MA, Colau B, Suzich J, Losonksy G, Martin MT, Dubin G, Wettendorff MA. Enhanced humoral and memory B cellular immunity using HPV16/18 L1 VLP vaccine formulated with the MPL/aluminium salt combination (AS04) compared to aluminium salt only. Vaccine. 2006 Aug 14;24(33-34):5937-49. doi: 10.1016/j.vaccine.2006.06.005. Epub 2006 Jun 19. PMID 16828940
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 580299/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 580299/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 580299/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 580299/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 580299/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 580299/005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register